CLINICAL TRIAL: NCT00809614
Title: Randomized, Double-blind Placebo-controlled Multi-center Proof-of-concept Study to Assess the Efficacy of AIN457 in Patients With Psoriatic Arthritis
Brief Title: Efficacy of AIN457 in Adults (18-65 Years) With Psoriatic Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457A2206
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Results first posted 2015-11-13 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-10

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic arthritis; IgG1K monoclonal antibody; Interleukin -17A neutralizing
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AIN457 (2x 10mg/kg) (Experimental): Each patient received 10 mg/kg AIN457 intravenously, on Day 1 and Day 22.
  Interventions: Biological: AIN457
- Placebo (Placebo Comparator): Each patient received 10 mg/kg of matching placebo intravenously, on Day 1 and Day 22.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: AIN457 — The investigational drug, AIN457 50 mg lyophilizate vials was prepared by Novartis. Reconstitution of AIN457 with 1.2 mL SWFI produced a 47 mg/mL concentrate solution for infusion from which at least 1 mL was useable. The AIN457 concentrate was diluted in 5% glucose bags for infusion through a 0.2 micron in-line filter.
  Arms: AIN457 (2x 10mg/kg)
Biological: Placebo — Matching placebo to AIN457
  Arms: Placebo

SUMMARY:
This study is designed as a proof of concept of AIN457 in patients with psoriatic arthritis. The study will address the evaluation of the efficacy at 6 and up to 24 weeks after two doses of AIN457 10 mg/kg administered three weeks apart.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of psoriatic arthritis

Exclusion Criteria:

* Patients with arthritis or ankylosing spondyitis
* Drug-induced psoriasis
* Male or female patients who plan to conceive during the time course of the study, or for 6 months after the administration of the second dose.
* Participation in any clinical trial within 4 weeks prior to initial dosing or longer.
* Previous use of immunosuppressive agents eg cyclosporine, without the necessary wash-out period
* History of severe allergy to food or drugs
* Positive TB test. Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis, Principal Investigator — Novartis Investigator Site
Locations (9):
- Germany (4):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, München
- Netherlands (2):
  - Novartis Investigative Site, Amsterdamn, DE
  - Novartis Investigative Site, Meerssen, KR
- United Kingdom (3):
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, Newcastle upon Tyne

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 42 patients were planned and recruited. The patients were randomized to either AIN457 2x10 mg/kg or placebo in a ratio of 2:1. The total sample size of 42 included an additional 3 subjects to allow for drop-outs and/or incomplete data.
Period: Overall Study
Arm/Group | AIN457 (2x 10mg/kg) | Placebo
Started | 28 | 14
Pharmacokinetic Safety Set | 27 | 14
Pharmacodynamic (PD) Set | 24 | 13
Completed | 25 | 10
Not Completed | 3 | 4
Not completed — Lack of Efficacy | 2 | 3
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: All patients who received at least one dose of study drug were included in the safety and tolerability evaluation.
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457 (2x 10mg/kg) | Placebo | Total
Number analyzed (Participants) | 28 | 14 | 42
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.7 (11.3) | 47.6 (8.1) | 47.0 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 8 | 27
  Male | 9 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of ACR Responders Per Treatment at Week 6
Description: A participant was considered to be a responder according to the ACR20, 50 or 70 criteria if the participant had at least 20% 50% or 70% improvement in both the tender joint count and swollen joint count measures, and in at least 3 of the following 5 measures: patient's assessment of pain, patient's global assessment of disease activity, physician's global assessment of disease activity, Health Assessment Questionnaire (HAQ©) score, and/or C-reactive protein (CRP)
Time Frame: week 6
Population: For pharmacodynamic (PD) analysis set five patients were excluded due to protocol deviations.
Measure: Number; unit: Percentage of ACR responders
Arm/Group | AIN457 (2x 10mg/kg) | Placebo
Number analyzed (Participants) | 24 | 13
Percentage of ACR responders
  ACR20 responders | 39 | 23
  ACR50 responders | 17 | 8
  ACR70 responders | 9 | 0

2. Primary Outcome: Percentage of PsARC Responders Per Treatment at Week 6
Description: Psoriatic Arthritis Response Criteria (PsARC) includes measures of tender and swollen joint counts, patient's assessment of pain, physician's and patient's global assessment of disease activity
  A subject is defined as a PsARC responder if, and only if, they have an improvement in two of the following four factors (with at least one factor being a joint count) and no worsening in the remaining factors: 1) Patient global assessment (0-100 VAS scale, improvement defined as decrease of at least 20 units) 2) Physician global assessment (0-100 VAS scale, improvement defined as decrease of at least 20 units) 3) Tender 78-joint count (improvement defined as decrease of at least 30%) 4) Swollen 76-joint count (improvement defined as decrease of at least 30%)
Time Frame: week 6
Population: For pharmacodynamic (PD) analysis set five patients were excluded due to protocol deviations.
Measure: Number; unit: Percentage of PsARC responders
Arm/Group | AIN457 (2x 10mg/kg) | Placebo
Number analyzed (Participants) | 24 | 13
Percentage of PsARC responders | 43 | 38

3. Secondary Outcome: Percentage of Participants Who Achieved 20%, 50% or 70% Improvement as Measured by ACR Response Criteria
Description: as for outcome 1
Time Frame: Day 8 and 15, Weeks 6, 8, 12, 16 and 24
Population: For pharmacodynamic (PD) analysis set five patients were excluded due to protocoldeviations.
Measure: Number; unit: Percentage of particpants
Arm/Group | AIN457 (2x 10mg/kg) | Placebo
Number analyzed (Participants) | 24 | 13
Percentage of particpants
  Day 8 ACR20 responders | 17 | 8
  Day 8 ACR50 responders | 0 | 0
  Day 8 ACR70 responders | 0 | 0
  Day 15 ACR20 responders | 25 | 17
  Day 15 ACR50 responders | 13 | 0
  Day 15 ACR70 responders | 0 | 0
  Week 6 ACR20 responders | 39 | 23
  Week 6 ACR50 responders | 17 | 8
  Week 6 ACR70 responders | 9 | 0
  Week 8 ACR20 responders | 42 | 23
  Week 8 ACR50 responders | 29 | 8
  Week 8 ACR70 responders | 17 | 0
  Week 12 ACR20 responders | 39 | 15
  Week 12 ACR50 responders | 22 | 8
  Week 12 ACR70 responders | 9 | 8
  Week 16 ACR20 responders | 41 | 27
  Week 16 ACR50 responders | 27 | 18
  Week 16 ACR70 responders | 18 | 9
  Week 24 ACR20 responders | 43 | 18
  Week 24 ACR50 responders | 17 | 9
  Week 24 ACR70 responders | 13 | 9

4. Secondary Outcome: Percentage of Participants Who Achieved PsARC Response
Description: responder" defined as 20% or more improvement in at least 4 of 6 criteria: 1) swollen joint count, 2) tender joint count, 3) morning stiffness duration (low back), 4) current low back pain, 5) current peripheral joint pain, 6) patient global assessment A subject is defined as a PsARC responder if, and only if, they have an improvement in two of the following four factors (with at least one factor being a joint count) and no worsening in the remaining factors: 1) Patient global assessment (0-100 VAS scale, improvement defined as decrease of at least 20 units) 2) Physician global assessment (0-100 VAS scale, improvement defined as decrease of at least 20 units) 3) Tender 78-joint count (improvement defined as decrease of at least 30%) 4) Swollen 76-joint count (improvement defined as decrease of at least 30%)
Time Frame: Day 8 and 15, Weeks 6, 8, 12, 16 and 24
Population: For pharmacodynamic (PD) analysis set five patients were excluded due to protocol deviations.
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 (2x 10mg/kg) | Placebo
Number analyzed (Participants) | 24 | 13
Percentage of participants
  Day 8 | 27 | 23
  Day 15 | 33 | 15
  Week 6 | 43 | 38
  Week 8 | 52 | 38
  Week 12 | 52 | 15
  Week 16 | 55 | 36
  Week 24 | 50 | 36

5. Secondary Outcome: Mastricht Ankylosing Spondylitis Enthesis Score (MASES) Over Time Per Treatment
Description: The MASES included assessments of 13 sites. Enthesitis sites included in the MASES index are: 1st costochondral, 7th costochondral, posterior superior iliac spine, anterior superior iliac spine, iliac crest (all above was assessed bilaterally), 5th lumbar spinous process, proximal Achilles (bilateral). The MASES score is defined as the total number of painful MASES entheses. The score was derived as the sum of the 13 scores divided by 3 and the total range is 0 (no tenderness) to 13 (severe tenderness).
Time Frame: Baseline and Day 8, 15 and weeks 6, 8, 12, 16 and 24
Population: For pharmacodynamic (PD) analysis set five patients were excluded due to protocol deviations
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AIN457 (2x 10mg/kg) | Placebo
Number analyzed (Participants) | 24 | 13
Units on a scale
  Baseline (n=24,13) | 3.0 (4.12) | 3.4 (2.33)
  Day 8 (n=23,13) | 2.6 (4.30) | 2.7 (2.59)
  Day 15 (24,13) | 2.9 (4.81) | 2.8 (3.42)
  Week 6 (n=23,11) | 2.6 (4.68) | 2.8 (3.34)
  Week 8 (n=22,11) | 2.7 (4.14) | 2.6 (3.32)
  Week 12 (n=20,11) | 2.4 (4.06) | 2.5 (2.62)
  Week 16 (n=19,9) | 2.6 (4.78) | 2.0 (2.40)
  Week 24 (n=23,11) | 1.6 (3.88) | 2.7 (3.32)

6. Secondary Outcome: Psoriatic Area and Severity Index (PASI) Score in Patients Over Time Per Treatment
Description: The PASI assessed the extent of psoriasis on four body surface areas (head, trunk and upper and lower limbs) and the degree of plaque erythema, scaling and thickness. The PASI score accounted for the extent of body surface area affected by the erythema, scaling and thickness, and the severity of these measures. The score ranged from 0 (no disease) to 72 (maximal disease).
Time Frame: Baseline, Day 8, 15 and weeks 6, 8, 12, 16, 20 and 24
Population: For pharmacodynamic (PD) analysis set five patients were excluded due to protocol deviations
Measure: Mean (Standard Deviation); unit: Unit on a Scale
Arm/Group | AIN457 (2x 10mg/kg) | Placebo
Number analyzed (Participants) | 24 | 13
Unit on a Scale
  Baseline (n=24,13) | 3.5 (4.20) | 2.4 (2.13)
  Week 6 (n=23,11) | 1.0 (1.5) | 3.10 (4.94)
  Week 12 (n=20,11) | 0.71 (1.12) | 3.3 (5.90)
  Week 24 (n=23,11) | 1.2 (1.67) | 3.6 (5.39)
  Day 8 (n=23,13) | 2.2 (2.77) | 2.3 (2.34)
  Day 15 (n=24,13) | 2.2 (2.92) | 2.2 (2.79)
  Week 8 (n=22,11) | 0.91 (1.43) | 3.5 (6.57)
  Week 16 (n=19,9) | 0.91 (1.25) | 4.2 (8.13)
  Week 20 (n=19,8) | 0.85 (1.36) | 3.84 (6.66)

7. Secondary Outcome: SpA Research Consortium of Canada (SPARCC) Score Score in Patients Over Time Per Treatment
Description: SPARCC evaluated 18 enthesis sites: medial and lateral epicondyle humerus, supraspinatus insertion, proximal Achilles, greater trochanter, medial and lateral condyl femur, insertion of plantar fascia, quadriceps insertion of patella, inferior pole of patella, and tibial tubercle. SPARCC enthesis index is defined as the total number of painful entheses assessed at the SPARCC sites. Total SI joint scores could range from 0 to 78, with a higher score indicating more signs of disease.
Time Frame: Baseline, Day 8, 15 and weeks 6, 8, 12, 16 and 24
Population: For pharmacodynamic (PD) analysis set five patients were excluded due to protocol deviations
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | AIN457 (2x 10mg/kg) | Placebo
Number analyzed (Participants) | 24 | 13
Unit on a scale
  Baseline (n=24,13) | 4.42 (5.055) | 6.08 (4.406)
  Week 6 (n=23,11) | 3.65 (5.515) | 4.27 (4.880)
  Week 12 (n=20,11) | 4.10 (5.428) | 5.27 (4.452)
  Week 24 (n=23,11) | 3.22 (5.161) | 4.36 (4.884)
  Day 8 (23,13) | 3.78 (5.054) | 4.08 (3.840)
  Day 15 (n=24,13) | 4.50 (6.400) | 4.15 (4.356)
  Week 8 (n=22,11) | 4.45 (4.993) | 4.00 (4.266)
  Week 16 (n=19,9) | 3.86 (5.844) | 3.67 (3.354)

8. Secondary Outcome: Leeds Dactylitis Instrument (LDI) Score in Patients Over Time Per Treatment
Description: The LDI basic measured the ratio of the circumference of the affected digit to the circumference of the digit on the opposite hand or foot, using a minimum difference of 10% to define a dactylitic digit. The ratio of circumference was multiplied by a tenderness score, using a modification of LDI which was a binary score (1 for tender, 0 for non-tender). If both sides were considered involved, the number was compared to data provided in a table. This modification was referred to as LDI basic and was applied in this study. The LDI required a tool to measure digital circumference and this tool was provided to the centers.
Time Frame: Baseline, Day 8, 15 and weeks 6, 8, 12, 16 and 24
Population: Only participants from the pharmacodynamic (PD) analysis set, who had available scores at each given time point, were analyzed for that time point. The PD analysis set included all patients with evaluable PD data with no protocol deviations that impacted PD data analysis.
Measure: Mean (Standard Deviation); unit: total score
Arm/Group | AIN457 (2x 10mg/kg) | Placebo
Number analyzed (Participants) | 6 | 7
total score
  Baseline (n=6,5) | 2.74 (2.32) | 1.56 (2.35)
  Week 6 (n=4,5) | 2.92 (2.37) | 2.14 (2.56)
  Week 12 (n=3,6) | 2.52 (1.57) | 0.73 (0.58)
  Week 24 (n=2,6) | 3.08 (1.54) | 1.88 (2.19)
  Day 8 (n=5,5) | 2.65 (1.60) | 1.32 (0.94)
  Day 15 (n=4,5) | 2.67 (2.61) | 1.72 (2.25)
  Week 8 (n=3,5) | 2.96 (1.03) | 1.54 (2.35)
  Week 16 (n=3,4) | 2.65 (1.82) | 2.08 (2.40)

9. Secondary Outcome: Disease Activity Score 28 (DA28) in Patients Over Time Per Treatment
Description: The Disease Activity Score (DAS) is a combined index to measure disease activity in arthritic patients. DAS28 is determined using the following variables: 28-joint counts (tender28 and swollen28), CRP, and the participant's general health (GH) Based on the patients global disease activity measured on a Visual Analogue Scale (VAS) of 100 mm (0 - 100). Using the data from these variables, DAS28 is calculated using the following formula: DAS28 = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.36*ln(CRP+1) + 0.014*GH + 0.96. The calculation results in a DAS28 score from 0 to 10 indicating the current activity of the rheumatoid arthritis of the patient. A DAS28 above 5.1 means high disease activity whereas a DAS28 below 3.2 indicates low disease activity. Remission is achieved by a DAS28 lower than 2.6.
Time Frame: Baseline, day 8, 15 and weeks 6, 8, 12, 16 and 24
Population: For pharmacodynamic (PD) analysis set five patients were excluded due to protocol deviations
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AIN457 (2x 10mg/kg) | Placebo
Number analyzed (Participants) | 24 | 13
Units on a scale
  Baseline (n=24,13) | 4.84 (1.21) | 4.76 (1.19)
  Week 6 (n=28,12) | 3.94 (1.47) | 4.20 (1.20)
  Week 12 (n=23,11) | 3.62 (1.42) | 4.36 (1.41)
  Week 24 (n=23,11) | 3.84 (1.30) | 4.28 (1.40)
  Day 8 (22,12) | 4.19 (1.27) | 4.43 (1.27)
  Day 15 (24,13) | 4.09 (1.26) | 4.35 (1.05)
  Week 8 (n=22,10) | 3.66 (1.65) | 4.64 (1.22)
  Week 16 (n=18,9) | 3.54 (1.48) | 3.83 (1.58)

10. Secondary Outcome: Pharmacokinetic (PK) of AIN457: Time to Reach the Maximum Concentration After Drug Administration (Tmax)
Description: On dosing days (Day 1 and Day 22) samples were taken at pre-dose (0 h), 2, 3, 4, 24. After the first infusion samples were taken at Day 8 and Day 15. After the second infusion samples were taken at Day 29, Day 43, Day 57, Day 71, Day 85, Day 113, Day 141, Day 169.
Time Frame: Day 1 till end of the study (169)
Population: Only patients who recieved active drug with evaluable pharmacokinetic ( PK) parameter data and no protocol deviation that impacted PK were included in the PK data analysis set
Measure: Median (Full Range); unit: Day
Arm/Group | AIN457 (2x 10mg/kg)
Number analyzed (Participants) | 27
Day | 21.0 [0.0833 to 23.1]

11. Secondary Outcome: Pharmacokinetic (PK) of AIN457: Clearance of AIN457 After Single Dose Administration
Description: as for outcome 10
Time Frame: Day 1 till end of the study (169)
Population: Only patients who recieved active drug with evaluable pharmacokinetic (PK) parameter data and no protocol deviation that impacted PK were included in the PK data analysis set
Measure: Mean (Standard Deviation); unit: Liters/day
Arm/Group | AIN457 (2x 10mg/kg)
Number analyzed (Participants) | 24
Liters/day | 0.161 (0.0535) [0.0833 to 23.1]

12. Secondary Outcome: Pharmacokinetic (PK) of AIN457: Terminal Elimination Half-life (T1/2)
Description: as for outcome 10
Time Frame: Day 1 till end of the study (169)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: day
Arm/Group | AIN457 (2x 10mg/kg)
Number analyzed (Participants) | 24
day | 29.8 (4.74) [0.0833 to 23.1]

13. Secondary Outcome: Pharmacokinetic (PK) of AIN457: Observed Maximum Serum Concentration Following Drug Administration (Cmax)
Description: as for outcome 10
Time Frame: Day 1 till end of the study (169)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | AIN457 (2x 10mg/kg)
Number analyzed (Participants) | 27
ug/mL | 424 (113) [0.0833 to 23.1]

14. Secondary Outcome: PK of AIN457: Area Under the Serum Concentration-time Curve From Time Zero to the Time of Last Quantifiable Concentration (AUClast), Area Under the Serum Concentration-time Curve From Time Zero to (AUCinf)
Description: as for outcome 10
Time Frame: Day 1 till end of the study (169)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | AIN457 (2x 10mg/kg)
Number analyzed (Participants) | 24
day*ug/mL
  AUClast | 12300 (2240) [0.0833 to 23.1]
  AUCinf | 12600 (2320)

15. Secondary Outcome: Pharmacokinetic (PK) of AIN457: Volume of Distribution During the Terminal Phase Following Intravenous Elimination (Vz)
Description: as for outcome 10
Time Frame: Day 1 till end of the study (169)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | AIN457 (2x 10mg/kg)
Number analyzed (Participants) | 24
Liters | 6.81 (2.17) [0.0833 to 23.1]

ADVERSE EVENTS:
Description: The Safety Set includes all subjects who received at least one dose of study medication
Groups:
- AIN457 2x10mg/kg: Each patient received 10 mg/kg AIN457 intravenously, on Day 1 and Day 22.
Arm/Group | AIN457 2x10mg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 4/28 | 1/14
Other Adverse Events (participants affected / at risk) | 23/28 | 11/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 2x10mg/kg (N=28) | Placebo (N=14)
Cellulitis (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 2x10mg/kg (N=28) | Placebo (N=14)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 3
Conjunctivitis (Eye disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 4 | 1
Periodontitis (Gastrointestinal disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 3 | 0
Pyrexia (General disorders) | 1 | 1
Bronchitis (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 7 | 5
Oral herpes (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 1
Neutrophil count decreased (Investigations) | 2 | 0
Red blood cell sedimentation rate increased (Investigations) | 2 | 1
White blood cell count decreased (Investigations) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Dizziness (Nervous system disorders) | 4 | 0
Headache (Nervous system disorders) | 6 | 1
Haematuria (Renal and urinary disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1
Haematoma (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety